CLINICAL TRIAL: NCT05810168
Title: Randomised Trial of Traditional Dietary Advice Versus a Low FODMAP Diet in Postprandial Functional Dyspepsia
Brief Title: Traditional Dietary Advice Versus Low FODMAP Diet in Postprandial Functional Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STH20655c
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Dyspepsia; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Dyspepsia; Gastrointestinal Diseases | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Traditional Dietary Advice (Active Comparator): Recommended to eat smaller, regular meals and reduce the intake of caffeine/alcohol/fizzy drinks, fatty/processed/spicy foods, and fibre
  Interventions: Other: Dietary modifications
- Low FODMAP diet (Active Comparator): FODMAPs are fermentable carbohydrates that increase intestinal water and gas production that, in those with visceral hypersensitivity, induces gastrointestinal symptoms. The low FODMAP diet therefore excludes fermentable carbohydrates, which are present in wheat-based products, many fruits/vegetables, pulses, beans, dairy, and sweeteners.
  Interventions: Other: Dietary modifications

INTERVENTIONS:
Other: Dietary modifications — TDA and low FODMAP diet

SUMMARY:
Functional dyspepsia is common, affecting 7.2% of the global population, and associated with substantial health impairment. Almost 80% of patients with functional dyspepsia report meal-related symptoms and are classified as having the postprandial distress syndrome (PDS) variant. However, studies evaluating dietary modifications in PDS are sparse.

The investigators will perform a randomised trial evaluating traditional dietary advice (TDA) vs. a diet low in fermentable fermentable oligo-, di-, mono- saccharides and polyols (low FODMAP diet) in PDS.

70 patients with PDS will be randomly assigned TDA or a low FODMAP diet. The TDA group will be recommended to eat small, regular meals and reduce the intake of caffeine/alcohol/fizzy drinks, fatty/processed/spicy foods, and fibre. The low FODMAP diet group will be advised to exclude fermentable carbohydrates, which are present in wheat-based products, many fruits/vegetables, pulses, beans, dairy, and sweeteners.

Questionnaires are to be completed during the 6-week trial, including self-reported adequate relief of dyspeptic symptoms, and the validated Leuven Postprandial Distress Scale (LPDS), Gastrointestinal Symptom Rating Scale, and Nepean Dyspepsia Quality of Life Index.

The primary endpoint to define clinical response will be evaluated over weeks 4-6 as >0.5-point reduction in the PDS subscale of the LPDS (calculated as the mean scores for early satiety, postprandial fullness, and upper abdominal bloating).

ELIGIBILITY:
Inclusion Criteria:

* Fulfil Rome IV symptoms criteria for postprandial functional dyspepsia
* Normal upper gastrointestinal endoscopy within last 3years
* Online access
* English literate

Exclusion Criteria:

* Organic gastrointestinal diseases (e.g. inflammatory bowel disease, GI cancer, coeliac disease)
* Major abdominal surgery (except laparoscopy, appendectomy, cholecystectomy)
* Documented H.pylori in the last 3 months
* History of eating disorders
* Body mass index <20
* Current dietary interventions
* Current use of opioids or anti-inflammatory drugs
* Severe systemic disease (e.g. cardiac, renal, respiratory) necessitating frequent medical consultations)
* Pregnant
* Diabetes mellitus
* Scleroderma
* Memory impairment

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of clinical responders between traditional dietary advice vs. a Low FODMAP diet on the leuven postprandial distress scale (LPDS) | 6 weeks
  The Leuven Postprandial Distress Scale (LPDS) assesses the severity of 8 upper gastrointestinal symptoms scored from 0 (none) to 4 (very severe). A difference of 0.5 from baseline for the cardinal PDS symptoms (average of first 3 questions) will be used as a cut-off to determine clinical response by comparing average pre-treatment scores with the average score during weeks 4-6.

SECONDARY OUTCOMES:
Proportion of clinical responders between traditional dietary advice vs. a low FODMAP diet | 6 weeks
  Self-reported adequate relief of dyspeptic symptoms as a binary answer (yes or no). A responder will be defined if ≥50% adequate relief of dyspeptic symptoms during weeks 4-6
Changes in Gastrointestinal Symptom Rating Irritable Bowel syndrome Scale | 6 weeks
  The validated Gastrointestinal Symptom Rating Scale assesses the symptoms of irritable bowel syndrome, depicting problems with satiety, abdominal pain, diarrhoea, constipation and bloating. Higher scores represent greater symptom severity. Change in scores will be compared within- and between- groups.
Changes in Napean Dyspepsia-related Quality of Life Index | 6 weeks
  The Napean Dyspepsia Scale is a validated questionnaire assessing dyspepsia-related quality of life syndrome, with higher scores representing worse quality of life. Change in scores will be compared within- and between- groups
Changes in Hospital Anxiety and Depression scale | 6 weeks
  The Hospital Anxiety and Depression Scale is a validated questionnaire assessing mood, with higher scores representing worse mood. Change in scores will be compared within- and between- groups
Changes in Somatic Symptom reporting | 6 weeks
  The validated patient health questionnaire-12 assess extra-intestinal somatic symptoms, with higher scores representing greater somatic symptom severity. Change in scores will be compared within- and between- groups
Changes in nutritional intake | 6 weeks
  The Comprehensive Nutritional Assessment Questionnaire assesses macronutrient and micronutrient intake, FODMAPs, fibre, starch, glycaemic index/load. Change in scores will be compared within- and between- groups

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No